CLINICAL TRIAL: NCT04977518
Title: Study of the Clinical Presentations, Treatment and Outcomes of Infective Endocarditis Patients in a Tertiary Hospital in East China
Brief Title: Characteristics of Infective Endocarditis in East China
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-046
Record Dates: First submitted 2021-07-13; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2016-03

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed during 2008-2011: Patients diagnosed with definite and probable infective endocarditis defined according to the modified Duke clinical criteria during 2008-2011
  Interventions: Other: no intervention
- Patients diagnosed during 2012-2015: Patients diagnosed with definite and probable infective endocarditis defined according to the modified Duke clinical criteria during 2012-2015
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This was a retrospective observational study of consecutive cases of definite or possible infective endocarditis (IE) as per the modified Duke criteria between January 2008 and December 2015, which was performed at the Second Affiliated Hospital of Zhejiang University, School of medicine (SAHZU), a tertiary care referral hospital located in East China.

DETAILED DESCRIPTION:
Infective endocarditis (IE) is a rare but life-threatening serious disease that still has a high mortality, even in developed countries. The objective of this study was to evaluate the clinical presentations, treatment and outcomes of IE patients in a tertiary hospital in East China over an 8-year period. This was a retrospective observational study of consecutive cases of definite or possible IE as per the modified Duke criteria between January 2008 and December 2015.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of infective endocarditis.

Exclusion Criteria:

* Patients did not meet the modified Duke criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a clinical diagnosis of infective endocarditis between January 2008 and December 2015 in a tertiary hospital located in the East China
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
Complications (neurological events, systemic embolism, and congestive heart failure) of infective endocarditis | During the hospitalization, average of 1 months
  1. A neurological event was defined as symptomatic or asymptomatic stroke, hemorrhage, or encephalopathy.
  2. Systemic embolization was defined as an embolic event outside of the central nervous system.
  3. Congestive heart failure was defined as with class III, or IV heart failure and an ejection fraction of 40% or less.
Mortality | During the hospitalization, average of 1 months
  Patients dead or moribund before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Huimin Xu, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: No
Data shared by published papers.